CLINICAL TRIAL: NCT04271306
Title: A Phase Ib Age De-escalation and Dose Escalation Open Label Clinical Trial of the Safety, Immunogenicity and ex Vivo Efficacy of a Candidate Malaria Vaccine Pfs25-IMX313/Matrix-M Administered Intramuscularly in Healthy Adults and Young Children in Tanzania.
Brief Title: Safety, Immunogenicity and ex Vivo Efficacy of Pfs25-IMX313/Matrix-M in Healthy Volunteers in Bagamoyo, Tanzania.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to significant delays in receiving local regulatory approval to extend the shelf-life of the IMP.
Sponsor: University of Oxford (Other)
Collaborators: Ifakara Health Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAC082
Record Dates: First submitted 2020-02-07; First posted 2020-02-17 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Malaria,Falciparum
Keywords: Vaccine
MeSH Terms: conditions — Malaria, Falciparum | interventions — Matrix-M

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Groups 1A & 1B (Experimental): Volunteers aged 18-45 years will receive doses of Pfs25-IMX313 (10µg)/Matrix-M (50µg) intramuscularly at months 0, 1 and 2
  Interventions: Biological: Pfs25-IMX313 (10ug)/Matrix-M (50ug)
- Groups 2A & 2B (Experimental): Volunteers aged 18-45 years will receive doses of Pfs25-IMX313 (50µg)/Matrix-M (50µg) intramuscularly at months 0, 1 and 2
  Interventions: Biological: Pfs25-IMX313 (50ug)/Matrix-M (50ug)
- Groups 3A & 3B (Experimental): Volunteers aged 5-12 years will receive doses of Pfs25-IMX313 (10µg)/Matrix-M (50µg) intramuscularly at months 0, 1 and 2
  Interventions: Biological: Pfs25-IMX313 (10ug)/Matrix-M (50ug)
- Group 3C (Experimental): Volunteers aged 5-12 years will receive doses of Pfs25-IMX313 (10µg)/Matrix-M (50µg) intramuscularly at months 0, 1 and 6.5
  Interventions: Biological: Pfs25-IMX313 (10ug)/Matrix-M (50ug)
- Groups 4A & 4B (Experimental): Volunteers aged 5-12 years will receive doses of Pfs25-IMX313 (50µg)/Matrix-M (50µg) intramuscularly at months 0, 1 and 6.5
  Interventions: Biological: Pfs25-IMX313 (50ug)/Matrix-M (50ug)
- Group 4C (Experimental): Volunteers aged 5-12 years will receive doses of Pfs25-IMX313 (50µg)/Matrix-M (50µg) intramuscularly at months 0 and 1 and a dose of Pfs25-IMX313 (10µg)/Matrix-M (50µg) intramuscularly at month 6.5
  Interventions: Biological: Pfs25-IMX313 (50ug)/Matrix-M (50ug) & Pfs25-IMX313 (10ug)/Matrix-M (50ug)

INTERVENTIONS:
Biological: Pfs25-IMX313 (10ug)/Matrix-M (50ug) — 3 doses of Pfs25-IMX313/Matrix-M at Pfs25-IMX313(10µg)/Matrix-M (50µg)
  Arms: Group 3C; Groups 1A & 1B; Groups 3A & 3B
Biological: Pfs25-IMX313 (50ug)/Matrix-M (50ug) — 3 doses of Pfs25-IMX313/Matrix-M at Pfs25-IMX313(50µg)/ Matrix-M (50µg)
  Arms: Groups 2A & 2B; Groups 4A & 4B
Biological: Pfs25-IMX313 (50ug)/Matrix-M (50ug) & Pfs25-IMX313 (10ug)/Matrix-M (50ug) — 2 doses of Pfs25-IMX313/Matrix-M at Pfs25-IMX313(50µg)/ Matrix-M (50µg) followed by one at Pfs25-IMX313(10µg)/Matrix-M (50µg)
  Arms: Group 4C

SUMMARY:
A phase Ib age de-escalation and dose escalation open label clinical trial of the safety, immunogenicity and ex-vivo efficacy of a candidate malaria vaccine Pfs25-IMX313/Matrix-M administered intramuscularly in healthy adults and young children in Tanzania

DETAILED DESCRIPTION:
This study aims to evaluate safety, immunogenicity, and transmission blocking activity of Pfs25IMX313-Matrix-M in healthy Tanzanian adults and children naturally exposed to malaria in Bagamoyo district, Tanzania. The study will enrol 45 volunteers comprising of 13 adults (18-45 years) and 32 children (5-12 years).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult aged 18 to 45 years or children aged 5-12 years.
2. Planned long-term (at least 30 months from the date of recruitment) or permanent residence in Bagamoyo town.
3. Adults with a Body Mass Index (BMI) 18 to 30 Kg/m2; or children (5-12 years) with the BMI between 13 and 25 Kg/m2.
4. Able and willing (in the Investigator's opinion) to comply with all study requirements.
5. Agreement to refrain from blood donation for the duration of the study
6. Written informed consent to participate in the trial.
7. Women only: Must practice continuous effective contraception* for the duration of the study.

Exclusion Criteria:

1. Use of immunoglobulins or blood products (e.g., blood transfusion) at any time in the past.
2. Receipt of any vaccine in the 14 days preceding enrolment, or planned receipt of any other vaccine within 14 days following each vaccination.
3. Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period.
4. Concurrent involvement in another clinical trial or planned involvement during the study period
5. Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data, as assessed by the Investigator
6. Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
7. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine (e.g. egg products)
8. Any history of anaphylaxis in reaction to vaccinations
9. Pregnancy, lactation or intention to become pregnant during the study.
10. History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
11. History of serious psychiatric condition that may affect participation in the study.
12. Any other serious chronic illness requiring hospital specialist supervision.
13. Suspected or known injecting drug abuse in the 5 years preceding enrolment.
14. Seropositive for hepatitis B surface antigen (HBsAg) or hepatitis C (HCV IgG).
15. Volunteers unable to be closely followed for social, geographic or psychological reasons.
16. Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination. In the event of clinically significant abnormal test results, confirmatory repeat tests will be requested. Procedures for identifying laboratory values meeting exclusion criteria will be described in a study specific SOP.
17. Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Ages: 5 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
Determine the safety of Pfs25IMX313-Matrix-M in healthy Tanzanian adults and children naturally exposed to malaria. | Assessment of solicited symptoms in the first 7 days post vaccination
  Occurrence of solicited symptoms after each vaccination during a 7-day surveillance period (day of vaccination and days 1, 2, 3 and 7 after vaccination).
Determine the safety of Pfs25IMX313-Matrix-M in healthy Tanzanian adults and children naturally exposed to malaria. | Assessment of unsolicited symptoms in the first 30 days post vaccination
  Occurrence of unsolicited symptoms after each vaccination during a 30-day surveillance period (day of vaccination and 30 subsequent days).
Determine the safety of Pfs25IMX313-Matrix-M in healthy Tanzanian adults and children naturally exposed to malaria. | Assessment of SAEs until the end of the study (approx 2 years)
  Occurrence of serious adverse events throughout the study period.

SECONDARY OUTCOMES:
Determine the Pfs25 specific antibody responses following immunization with different vaccination regimens in healthy Tanzanian adults and children. | Duration of the study (approx 2 years)
  Pfs25 antibody levels elicited by Pfs25IMX313-Matrix-M as measured by ELISA at each time point where serology samples are analysed.
Determine the transmission blocking activity of Pfs25 specific antibodies elicited by the different vaccination regimens in healthy Tanzanian adults and children using Standard Membrane Feeding Assay (SMFA) and Direct Membrane feeding assay (DMFA). | Duration of the study (approx 2 years)
  Transmission blocking activity (TBA) of induced antibody as measured in standard membrane feeding assays (SMFA) and Direct Membrane feeding assays (DMFA).
Determine the transmission blocking activity of Pfs25 specific antibodies elicited by the different vaccination regimens in healthy Tanzanian adults and children using Standard Membrane Feeding Assay (SMFA) and Direct Membrane feeding assay (DMFA). | Duration of the study (approx 2 years)
  Correlation of TBA with antibody levels at each time point where the membrane feeding assays are conducted.
Select the best vaccination regimen based on the peak Pfs25 specific antibodies after final immunization, their duration and transmission blocking activity by standard membrane feeding assay (SMFA) and direct membrane feeding assay (DMFA). | Duration of the study (approx 2 years)
  The vaccination schedule that lead to the highest peak and duration of anti-Pfs25 antibody response post vaccination, and the highest transmission blocking activity (TBA) as measured by standard membrane feeding assay (SMFA) and direct membrane feeding assay (DMFA).

CONTACTS AND LOCATIONS:
Overall Officials: Angela Minassian, Principal Investigator — University of Oxford
Locations (1):
- Ifakara Health Institute Clinical Trial Facility, Bagamoyo, Tanzania